CLINICAL TRIAL: NCT00128076
Title: All-Arthroscopic Versus Mini-Open Repair of Small or Moderate Rotator Cuff Tears
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Joy MacDermid, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCT-82335
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Shoulder Pain; Rotator Cuff Tear
Keywords: shoulder surgery; rotator cuff; arthroscopic repair; mini-open repair
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): All-arthroscopic repair
  Interventions: Procedure: All-Arthroscopic repair
- 2 (Active Comparator): Mini-open repair
  Interventions: Procedure: Mini-open repair

INTERVENTIONS:
Procedure: All-Arthroscopic repair — joint techniques and repair are both performed entirely through the arthroscope
  Arms: 1
Procedure: Mini-open repair — repair is performed though a small incision and the arthroscope can be used to address problems within the joint (as per traditional diagnostic procedures)
  Arms: 2

SUMMARY:
This study will compare two different surgical techniques for repairing a tear in the muscles of the shoulder (rotator cuff). The investigators will determine whether an arthroscopic or mini-open technique provides better quality of life and repair integrity.

DETAILED DESCRIPTION:
Background:

Rotator cuff tears are the most common source of shoulder pain and disability. Only poor quality studies have compared mini-open to arthroscopic repair, leaving surgeons with inadequate evidence to support optimal, minimally-invasive repair.

Methods/Design:

This randomized, multi-centre, national trial will determine whether an arthroscopic or mini-open repair provides better quality of life for patients with small or moderate sized rotator cuff tears. A national consensus meeting of investigators in Joints Orthopaedic Initiative for Shoulder Trials (JOINTS) identified this question as the top priority for shoulder surgeons across Canada. The primary outcome measure is a valid quality-of-life scale (Western Ontario Rotator Cuff (WORC) that addresses 5 domains of health affected by rotator cuff disease. Secondary outcomes will assess rotator cuff functionality (ROM, strength, constant score), secondary dimensions of health (general health status (SF-12) and work limitations) and repair integrity (MRI). Outcomes are measured at baseline, at 6 weeks, 3, 6, 12 and 24 months postoperatively by blinded research assistants and musculoskeletal radiologists. Patients (n=250) with small or medium-sized cuff tears identified by clinical examination and MRI who meet eligibility criteria will be recruited. This sample size will provide 80% power to detect (statistically) a clinically important difference of 20% in WORC scores between procedures after controlling for baseline WORC score ("=0.05). A central methods centre will manage randomization, data management and monitoring under supervision of experienced epidemiologists. Surgeons will participate in either conventional or expertise-based designs according to defined criteria, to avoid biases from differential surgeon expertise. Mini-open or all-arthroscopic repair procedures, will be performed according to a standardized protocol. Central Adjudication (of cases), Trial Oversight and Safety Committees will monitor trial conduct. The investigators will use an analysis of covariance (ANCOVA), where the baseline WORC score is used as a covariate, to compare the quality of life (WORC score) at 2-years post-operatively. As a secondary analysis the investigators will conduct the same statistical test but will include age and tear size as covariates with the baseline score. Enrollment will require 2 years and follow-up an additional 2-years.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will recruit patients with small or medium rotator cuff tears as determined by clinical examination and diagnostic imaging (magnetic resonance imaging [MRI]) prior to surgery.
* The full-thickness rotator cuff tears of supraspinatus and infraspinatus will be classified into 2 categories based on area of longest dimension.

  * SMALL= 0-1 cm;
  * MODERATE =1-3 cm.
* Definitive measurement of tear size will be made in surgery and used as a covariate in analysis. (JOINTS measurement protocol will be used)

Exclusion Criteria:

Pre-Operative Exclusion Criteria

* Evidence of major joint trauma, infection, avascular necrosis, chronic dislocation, inflammatory or degenerative glenohumeral arthropathy, frozen shoulder or previous surgery of the affected shoulder,
* Evidence of significant cuff arthropathy with superior humeral translation and acromial erosion diagnosed by x-ray or other investigations,
* Major medical illness (life expectancy less then 2 years or unacceptably high operative risk),
* Unable to speak or read English,
* Psychiatric illness that precludes informed consent,
* Unwilling to be followed for 2 years.

Intra-Operative Exclusion Criteria

* Large, massive or irreparable cuff tears, extending into the subscapularis or teres minor, which cannot be mobilized to the articular margin or repaired using one or both of the techniques (all arthroscopic or mini-open),
* Teres minor or subscapularis tears,
* Inelastic and immobile tendon, which cannot be advanced to articular margin,
* Co-existing labral pathologies requiring repair with sutures (superior labral anterior posterior [SLAP] II-IV), Bankart lesions requiring repair, partial tears of biceps (more than 60% of thickness) requiring tenodesis or release.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2006-08; Primary Completion 2014-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quality of life measure specific to rotator cuff disease (Western Ontario Rotator Cuff Questionnaire (WORC) | within 2 years

SECONDARY OUTCOMES:
SF-12 | within 2 years
Work Limitations Scale | within 2 years
Cuff integrity on imaging | within 1 year post-operative
Strength | within 2 years
Range of Motion | within 2 years
American Shoulder and Elbow Surgeons (ASES) shoulder scale | within 2 years
Shoulder and Pain Disability Index (SPADI) | Within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joy C MacDermid, PhD, Principal Investigator — McMaster University, University of Western Ontario
Locations (9):
- Canada (9):
  - University of Calgary Sport Medicine Centre, Calgary, Alberta
  - Walter Mackenzie Centre, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - PanAm Clinic, Winnipeg, Manitoba
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Fowler Kennedy Sports Medicine Clinic, London, Ontario
  - St. Joseph's Health Care London, London, Ontario
  - Orthopaedic and Arthritic Hospital, Toronto, Ontario

REFERENCES:
- [Background] MacDermid JC, Holtby R, Razmjou H, Bryant D; JOINTS Canada. All-arthroscopic versus mini-open repair of small or moderate-sized rotator cuff tears: a protocol for a randomized trial [NCT00128076]. BMC Musculoskelet Disord. 2006 Mar 10;7:25. doi: 10.1186/1471-2474-7-25. PMID 16529658
- [Derived] MacDermid JC, Bryant D, Holtby R, Razmjou H, Faber K; JOINTS Canada; Balyk R, Boorman R, Sheps D, McCormack R, Athwal G, Hollinshead R, Lo I, Bicknell R, Mohtadi N, Bouliane M, Glasgow D, Lebel ME, Lalani A, Moola FO, Litchfield R, Moro J, MacDonald P, Bergman JW, Bury J, Drosdowech D. Arthroscopic Versus Mini-open Rotator Cuff Repair: A Randomized Trial and Meta-analysis. Am J Sports Med. 2021 Oct;49(12):3184-3195. doi: 10.1177/03635465211038233. Epub 2021 Sep 15. PMID 34524031